CLINICAL TRIAL: NCT03410615
Title: Randomized Phase II Study of Cisplatin Plus Radiotherapy Versus Durvalumab Plus Radiotherapy Followed by Adjuvant Durvalumab Versus Durvalumab Plus Radiotherapy Followed by Adjuvant Tremelimumab and Durvalumab in Intermediate Risk HPV-Positive Locoregionally Advanced Oropharyngeal Squamous Cell Cancer (LA-OSCC)
Brief Title: Cisplatin + Radiotherapy vs Durvalumab + Radiotherapy Followed by Durvalumab vs Durvalumab + Radiotherapy Followed by Tremelimumab + Durvalumab in Intermediate-Risk HPV-Positive Oropharyngeal SCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN9
Record Dates: First submitted 2018-01-09; First posted 2018-01-25 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiation; Cisplatin; durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: This is a non-comparative, randomized, phase II study of cisplatin plus radiotherapy or durvalumab plus radiotherapy followed by adjuvant durvalumab or durvalumab plus radiotherapy followed by adjuvant tremelimumab and durvalumab in intermediate risk, HPV-positive, locoregionally advanced oropharyngeal squamous cell cancer (LA-OSCC) of the head and neck.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radiation/Cisplatin (Active Comparator): All patients will receive standard fractionation radiation therapy (RT) scheme: 70 Gy in 35 fractions over 7 weeks (i.e. 2 Gy per fraction)
  Cisplatin IV 100 mg/m2 days 1, 22, 43 concurrently with RT
  Interventions: Radiation: Radiation; Drug: Cisplatin
- Radiation/Durvalumab + Adjuvant Durvalumab (Experimental): All patients will receive standard fractionation radiation therapy (RT) scheme: 70 Gy in 35 fractions over 7 weeks (i.e. 2 Gy per fraction)
  Concurrent Phase: Durvalumab IV 1500 mg, days -7 and 22 (the second dose is given concurrently with RT).
  Adjuvant Phase (to start 4 weeks after completion of concurrent phase): Durvalumab IV 1500 mg q4 weekly for 6 doses.
  Interventions: Radiation: Radiation; Drug: Durvalumab
- Radiation/Durvalumab + Adjuvant Durvalumab/Tremelimumab (Experimental): ARM CLOSED TO ACCRUAL WITH AMENDMENT #1
  Interventions: Radiation: Radiation; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Radiation: Radiation — 70 Gy in 35 fractions over 7 weeks (i.e. 2 Gy per fraction)
Drug: Cisplatin — 100 mg/m2 days 1, 22, 43 concurrently with RT
  Arms: Radiation/Cisplatin
Drug: Durvalumab — Given in concurrent and adjuvant phase
  Arms: Radiation/Durvalumab + Adjuvant Durvalumab; Radiation/Durvalumab + Adjuvant Durvalumab/Tremelimumab
Drug: Tremelimumab — ARM CLOSED TO ACCRUAL - 2019
  Arms: Radiation/Durvalumab + Adjuvant Durvalumab/Tremelimumab

SUMMARY:
Sometimes, cancer patients receive an initial treatment, followed by additional treatment to lower the chance of cancer coming back. The standard or usual treatment for this type of disease is initially having radiation therapy at the same time as chemotherapy (with a drug called cisplatin), with no additional therapy afterwards

DETAILED DESCRIPTION:
This study is looking at whether a type of drug called durvalumab can be used with radiation during the initial treatment, (instead of cisplatin) and also afterwards as additional therapy. Durvalumab is an immunotherapy drug . It has been tested in many different types of cancers. Durvalumab works by allowing the immune system to detect the cancer and reactivate the immune response. This may help to slow down the growth of cancer or may cause cancer cells to die. Durvalumab has been shown to shrink tumours in animals. It has been studied in more than 5000 people, approved for use in other cancers and seems promising.

This clinical trial will also test another type of immunotherapy drug called tremelimumab, which would also be given as additional treatment. Tremelimumab works in a different way to durvalumab to enhance the immune system reaction against cancer cells and may improve the effect of durvalumab. Tremelimumab may also help slow the growth of the cancer cells or may cause cancer cells to die. It has been shown to shrink tumours in animals. Tremelimumab has been studied in over 1200 people, approved for use in other cancers and seems promising.

As of February 2019, tremelimumab will no longer be tested with new participants joining the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed (primary lesion or regional lymph nodes) squamous cell carcinoma of the oropharynx (OSCC) which is locoregionally advanced, intermediate risk and non-metastatic (M0) as defined by the following (UICC/AJCC 8th Edition staging)

  * T1-2 N1 (smoking ≥ 10 pack years);
  * T3 N0-N1 (smoking ≥ 10 pack years);
  * T1-3 N2 (any smoking hx).
* Human papillomavirus (HPV)-related as determined by positive p16 immunohistochemical staining on any tumour specimens. Positive p16 expression is defined as strong and diffuse nuclear and cytoplasmic staining in 70% or more of the tumour cells. Local testing is acceptable; testing will not be done centrally in real-time.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (see Appendix I) and a body weight of > 30 kg.
* The following radiological investigations must be done within 8 weeks of randomization:

  * CT or MRI of the neck (with PET-CT and head imaging as indicated);
  * CT chest or x-ray, other radiology tests as clinically indicated.
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method.
* Patient must consent to provision of, and investigator(s) must confirm location and commit to obtain a representation of formalin fixed paraffin block, of non-cytology tissue samples in order that the specific correlative mark assays may be conducted.
* Patient must consent to provision of samples of blood, saliva and oropharyngeal swab in order that the specific correlative marker assays may be conducted
* Patient is able (i.e. sufficiently fluent) and willing to complete the quality of life and health economics questionnaires in the languages provided.
* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre
* In accordance with CCTG policy, protocol treatment (cisplatin/RT or durvalumab) is to begin within 1 week of randomization.
* The patient is not receiving anti-cancer therapy in a concurrent clinical study testing new treatments or treatment strategies and the patient agrees not to participate in other clinical studies during their participation in this trial while on study treatment.
* Adequate normal organ and marrow function as defined below (must be done within 14 days prior to randomization): Absolute neutrophils - ≥ 1.5 x 10^9/L; Platelets ≥100 x 10^9; Hemoglobin ≥90 g/L; Bilirubin ≤ 1.5 x UNL; AST and ALT ≤2.5 x UNL; Creatine clearance ≥ 60 mL/min.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements
* Patients must be assessed by a radiation oncologist and medical oncologist and deemed suitable for study participation including administration of radiotherapy, cisplatin and durvalumab as outlined in the protocol.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumours curatively treated with no evidence of disease for ≥ 5 years.
* Current history of other non-OSCC malignancies of the head and neck.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab, or an anti-CTLA4, including tremelimumab.
* Any previous cisplatin or carboplatin chemotherapy.
* Any previous induction chemotherapy for current SCCHN.
* Any previous surgical treatment of the current cancer (except for a diagnostic biopsy) and no major surgery within 28 days prior to randomization.
* Any previous radiation to the head and neck region that would result in overlap of fields for the current study.
* History of allergic or hypersensitivity reactions to any study drug or their excipients.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 msec in screening ECG measured using standard institutional method or history of familial long QT syndrome.
* History of primary immunodeficiency, history of allogenic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization* or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction
* Current or prior use of immunosuppressive medication within 28 days of study entry, with the exceptions of intranasal and inhaled corticosteroids or systemic chronic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Corticosteroids used on study for anti-emetic purpose are allowed. Corticosteroids as premedication for hypersensitivity reactions (e.g. computed tomography [CT] scan premedication) are allowed.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease (controlled by diet alone) or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:
* Patients with vitiligo or alopecia;
* Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years);
* Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement;
* Any chronic skin condition that does not require systemic therapy.
* Patients with active or uncontrolled intercurrent illness including, but not limited to:

  * cardiac dysfunction (symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia);
  * active peptic ulcer disease or gastritis;
  * active bleeding diatheses;
  * psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent;
  * known history of previous clinical diagnosis of tuberculosis;
  * known active human immunodeficiency virus infection (positive HIV 1/2 antibodies); HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible;
  * known active hepatitis B infection (positive HBV surface antigen (HBsAg). Patients with a past or resolved HBV infection (defined as presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible;
  * known active hepatitis C infection. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline CT scan.
* Receipt of live attenuated vaccination (examples include, but are not limited to, vaccines for measles, mumps, and rubella, live attenuated influenza vaccine (nasal), chicken pox vaccine, oral polio vaccine, rotavirus vaccine, yellow fever vaccine, BCG vaccine, typhoid vaccine and typhus vaccine) within 30 days prior to randomization.
* Pregnant or lactating women
* Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
* Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
3 year event-free survival | 3 years
  Event-free survival (EFS), is defined as the time from randomization to the time when a failure event is observed. Failure is define by Local-regional progression or recurrence, Distant metastasis, Non-protocol RT, chemotherapy, Surgery or death.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Head and Neck Version (FACT-HN) score. | 6 years
  The FACT-H&N is a multidimensional, self-report QoL instrument specifically designed for use with head and neck cancer patients (1-3). It consists of 27 core items which assess patient function in four domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by 12 site specific items to assess for head and neck related symptoms.
  Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as an global QoL score. Higher scores represent better QoL.
Local regional failure | 6 years
  Locoregional control defined as time from randomization to the time of first documented local (primary site) or regional (lymph node) recurrence
Distant metastasis-free survival | 6 years
  Distant metastasis-free survival defined as time from randomization to the time of first documented distant metastasis or death from any cause
Overall survival | 6 years
  Overall Survival defined as time from randomization to the time of death from any cause
Cost-effectiveness of immunotherapy-based treatment arm vs standard of RT and cisplatin in patients with intermediate risk LA-OSC using the EQ-5D-5L | 6 years
Number and severity of adverse events | 6 years
Cost-utility will be used to abstract indirect costs at the end of RT and at 6 and 12 months post RT | 6 & 12 months
Lost productivity questionnaire will be used to abstract indirect costs at the end of RT and at 6 and 12 months post RT | 6 & 12 months
Incidence of second cancer | 6 years
PRO-CTCAE baseline, last week of treatment, 3 months, 6 months and 12, 24 and 36 months from the end of RT | 3, 6, 12, 24 and 36 months
Dysphagia: PSS-HN swallowing subscale at 36 months from the end of RT | 36 months
Dysphagia: using MDADI Global at 36 months from the end of RT | 36 months
Number and severity of radiation-related late toxicity at 3 months, 6 months and 1 year from the end of RT | 3 months, 6 months & 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anna Spreafico, Study Chair — UNH/Princess Margaret Cancer Centre, Toronto ON Canada; Khalil Sultanem, Study Chair — The Jewish General Hospital, Montreal QC, Canada
Locations (26):
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital of Antwerp, Edegem
  - University Hospital of Gent, Ghent
  - University Hospital Leuven, Leuven
  - Clinique St. Elizabeth, Namur
  - AZ Sint Augustinus, Wilrijk
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - The Jewish General Hospital, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Spain (5):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - University Hospital Vall dHebron, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - University Hospital Ramon y Cajal, Madrid
  - University Clinical Hospital of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No